CLINICAL TRIAL: NCT07104396
Title: Cogito: A Turnkey Solution for Rapidly Developing, Evaluating, Deploying, and Scaling Digital Therapeutics
Status: Recruiting | Type: Observational
Sponsor: Square2 Systems, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Grabinski, Principal Investigator, Square2 Systems, Inc.
Other Study IDs: 1R43DA060729-01 (NIH)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Substance Use Disorders (SUDs)
Keywords: digital therapeutics; substance use disorders; development platform
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cogito digital therapeutics development platform — Cogito will provide a turnkey solution for rapidly developing, evaluating, deploying, and scaling digital therapeutics for the prevention, treatment and/or management of any disease or disorder. This platform will allow researchers who are seeking to embed an evidence-based behavioral therapy into a digital delivery platform to do so via a drag and drop interface with no programming skills necessary. It will provide all the components for building a digital therapeutic for any health condition and population. Overall, Cogito offers great promise to markedly accelerate the pace and impact of science based digital therapeutics.

SUMMARY:
This is a research study to evaluate the usability of the Cogito digital therapeutics development platform.

The Cogito platform is designed to allow researchers who are seeking to embed an evidence-based behavioral therapy into a digital delivery platform to do so via a drag and drop interface with no programming skills necessary. It will provide the components for building a digital therapeutic for any health condition and population.

And in this initial study, the research team plans to examine the usability of Cogito in building a digital therapeutic for substance use disorders (SUDs).

DETAILED DESCRIPTION:
Each participant will be asked to:

* Complete an interactive tutorial describing what Cogito is and how to create a sample guide, sample activities, and a sample survey.
* Explore using the various Cogito processes by completing a "functionality scavenger hunt". In this scavenger hunt, participants will be walked through a series of activities to create new guides, activities and surveys.
* Complete surveys to provide feedback on participants' experience using Cogito

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years
* PhD and/or MD-level (or equivalent) scientists at academic institutions or digital health companies at the level of Post-doctoral Fellow or higher.
* Training or trained in substance use disorder (SUDs) research.
* Must state a specific interest in digital therapeutics for SUDs.

Exclusion Criteria:

* Those who do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research team will recruit 20 (> 18 years) clinical researchers/clinicians to utilize Cogito to provide feedback on its usability, utility, and likability and relevance as a development and hosting platform. Participants must be PhD and/or MD-level scientists at academic institutions or digital health companies at the level of Post-doctoral Fellow or higher. Participants must be trained/training in SUD research. Participants must state a specific interest in digital therapeutics for SUDs. The researchers expect participants will have interests ranging from developing novel behavioral digital therapies for SUDs to digital therapeutics that promote adherence to SUD medications to digital therapeutics for SUDs and co-occurring conditions to digital management tools which help individuals with care transitions.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | To be completed immediately after usability feedback session
  Each participant will be asked to complete the standardized 10-item System Usability Scale (SUS) to evaluate the usability of Cogito (e.g., "I think I would like to use this system frequently"), ranging from "strongly agree" to "strongly disagree".

SECONDARY OUTCOMES:
Visual Analog Scales | To be completed immediately after usability feedback session
  100 mm Visual Analog measures, ranging from "Not at All" anchored at 0 to "Very" anchored at 100 for each question, with every question worded positively to assess how (1) easy to use, (2) understandable, (3) likable, (4) useful (5) relevant they found the Cogito development functionality in each stage of the scavenger hunt as well as (6) how likely they would be to use Cogito as a digital therapeutics development and hosting platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Square 2 Systems, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided